CLINICAL TRIAL: NCT03878862
Title: Surgical Treatment of Massive and Irreparable Rotator Cuff Tears
Brief Title: Surgical Management of Irreparable RC Tears
Status: Recruiting | Type: Observational
Sponsor: Panam Clinic (Other)
Collaborators: Pan Am Clinic (Other)
Responsible Party: Principal Investigator, Peter MacDonald, Orthopaedic surgeon, Panam Clinic
Other Study IDs: H2018:135
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary goal will be to compare the early postoperative recovery outcomes and complications from a series of surgical treatments for massive or irreparable rotator cuff tears. The secondary goal will be to assess factors that impact the outcomes of these reconstructions for irreparable posterosuperior rotator cuff tears.

DETAILED DESCRIPTION:
Prospective, Non-Randomized Cohort Study The surgeons will decide which surgical reconstruction technique should be used to treat patients who have a massive (2+ tendons) or irreparable (Grade 3 or higher fatty infiltration into infraspinatus tendon) rotator cuff tear in the primary or revision setting. Surgical options include arthroscopic superior capsular reconstruction (SCR), arthroscopic assisted latissimus dorsi transfer (aaLDT), or arthroscopic assisted lower trapezius transfer (aaLTT), with arthroscopic biceps tendoesis/tenotomy as a control group.

Each patient will receive an X-ray and MRI to indicate reparable subscapularis tear, teres minor pathology, grade of muscle fatty infiltration, AHI, CSA, Hamada grade, and arthritis grade.

Patients will be assessed pre-operatively and again post-operatively at 6 weeks, 3 months, 6 months, 12 months, and 24 months to collect patient reported outcomes and complications. Assessments will include clinical and shoulder motion evaluations to gauge shoulder range of motion and pathology, as well as questionnaires that evaluate the patients shoulder mobility, ability, pain, and surgical satisfaction. Any adverse events post surgery will also be recorded at the defined assessment time intervals (6 wks, 3m, 6m, 12m, 24,m) and will specifically monitor temporary or permanent nerve injuries, hematomas, superficial and deep infections, recurrent moderate/severe pain, tendon or graft rupture, and humeral head superior migration.

Graphical comparisons will be made of the patient's recovery for each surgical technique as well as an analysis of patient specific factors based on their demographics forms which could influence the recovery curves.

ELIGIBILITY:
Inclusion Criteria:

* massive (2+ tendons) or irreparable (see below) rotator cuff tears in the primary or revision setting.

  * Definition of "irreparable": grade 3 or higher fatty infiltration into the infraspinatus

Exclusion criteria:

* Protected populations: prisoners, military, non-English speakers, age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting at the Pan Am Clinic to the contributing surgeons with an irreparable rotator cuff tear
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale for pain | 24-months
  10 cm scale with 0 = no pain and 10= extreme pain
Simple shoulder test | 24-months
  A validated score of items whereby patients indicate ability to perform or not with a lower score equal to worse outcomes. Maximum 12
American Shoulder and Elbow Score | 24-months
  Validated shoulder and elbow outcome with a maximum score of 30, with 0 being poor outcome and 30 being the most positive outcome
Veterans Rand - 12 | 24-months
  A validated general health survey with 0 as a poor outcome and 100 as a positive outcome.
Western Ontario Rotator Cuff score | 24-months
  A validated measure with 0 as a poor score and 100 as a positive score.

CONTACTS AND LOCATIONS:
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada